CLINICAL TRIAL: NCT04024254
Title: A Study of Serum Folate Levels in Patients With Treated With Olaparib.
Brief Title: A Study of Serum Folate Levels in Patients Treated With Olaparib
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Lydia Usha, Professor of Medicine, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18070604
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Breast Cancer; Folic Acid Deficiency
Keywords: ovarian cancer; breast cancer; olaparib; folic acid deficiency
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Folic Acid Deficiency | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Folic Acid supplementation (Experimental): Folic Acid supplement 1 mg by mouth daily
  Interventions: Drug: Folic Acid Tablet
- No Folic Acid Supplementation (No Intervention): No Folic Acid supplementation.

INTERVENTIONS:
Drug: Folic Acid Tablet — Folic Acid 1 mg by mouth daily
  Arms: Folic Acid supplementation

SUMMARY:
This is a study investigating folate deficiency (lack of folic acid in the blood) in patients who take the drug olaparib to treat their advanced ovarian or breast cancer.

DETAILED DESCRIPTION:
This is a study investigating folate deficiency (lack of folic acid in the blood) in patients who take the drug olaparib to treat their advanced ovarian or breast cancer. The primary goal of this study is to determine the frequency and timing of folate deficiency, and to learn more about whether giving folic acid supplementation (vitamin) will help delay or avoid deficiency in these patients. Deficiency can cause doctors to reduce or stop treatment with olaparib. In this case, patients are not getting the best treatment for their cancer due to the unwanted side effect.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed informed consent
* Female, post-menopausal, ≥18 years of age inclusive, at the time of signing the consent form
* Individuals who have ovarian cancer or breast cancer who are recommended to start olaparib
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:
* Haemoglobin ≥ 9 g/dL with no blood transfusion in the past 28 days
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
* Patients must have creatinine clearance estimated of ≥51 mL/min
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1).
* Patients must have a life expectancy ≥ 16 weeks.
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT and is suitable for repeated assessment.

Exclusion Criteria:

* Patients with folic acid deficiency, defined as folate <7 ng/mL, or those taking folic acid supplementation within 30 days of olaparib initiation.
* Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma. Patients with a history of localised triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with known active hepatitis (i.e. Hepatitis B or C).
* Any previous treatment with PARP inhibitor, including Olaparib.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).
* Participation in another clinical study with an investigational product administered in the last 1 month
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with a known hypersensitivity to folic acid or any of the excipients of the product.
* Involvement in the planning and/or conduct of the study
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Previous enrollment in the present study
* Breast feeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Usha, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol started in August 2020 and completed in August 2022. Patients were recruited from the Gynecologic Oncology and Breast Oncology clinics at a major medical center.
Pre-assignment Details: Patients who were planned to receive the PARP inhibitor, Olaparib for the treatment for Ovarian or Breast cancer were eligible for the study. After obtaining consent, screening activities included baseline blood work and physical exam. One of the ten subjects was excluded as it was revealed that she had received prior PARP inhibitor treatment on a blinded trial.
Groups:
- Folic Acid: Folic Acid supplement 1 mg by mouth daily
  Folic Acid Tablet: Folic Acid 1 mg by mouth daily
- No Supplementation: No Folate supplementation
Period: Overall Study
Arm/Group | Folic Acid | No Supplementation
Started | 2 | 7
Completed | 2 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Folic Acid Supplementation Group: Folic Acid supplement 1 mg by mouth daily
  Folic Acid Tablet: Folic Acid 1 mg by mouth daily
- Total: Total of all reporting groups
Arm/Group | Folic Acid Supplementation Group | No Supplementation | Total
Number analyzed (Participants) | 2 | 7 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 4 | 4
Age, Continuous [Median (Full Range); unit: years] — Age was listed as years of age and verified by date of birth found in the medical record.
  years | 49 [44 to 53] | 66 [43 to 89] | 64 [43 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 7 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All participants lived in the Chicagoland area in the United States.
  participants
    United States | 2 | 7 | 9
Folate levels at baseline [Mean (Full Range); unit: ng/mL] | 10.5 [7.3 to 13.7] | 18.6 [9.6 to 35.0] | 14.6 [7.3 to 35.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have Developed Folate Deficiency (Serum Folate Level < 7 ng/ml) on Olaparib
Description: The number of patients with ovarian and breast cancers who were treated with olaparib and developed folate deficiency was counted.
Time Frame: Serum folate levels were measured in each enrolled subject: at baseline, then every 2 weeks X 3 months, then monthly X 9 months. Accrual occurred over a 2-year period.
Measure: Count of Participants; unit: Participants
Groups:
- Folic Acid Supplementation Arm: Folic Acid supplement 1 mg by mouth daily
Arm/Group | Folic Acid Supplementation Arm | No Supplementation
Number analyzed (Participants) | 2 | 7
Participants | 2 | 6

2. Primary Outcome: Timing of Folate Deficiency Development
Description: The number of weeks between the beginning of olaparib treatment and the development of folate deficiency
Time Frame: From the beginning of olaparib treatment until the development of folate deficiency
Population: Only 6 subjects in the no folate supplementation arm developed folate deficiency.
Measure: Mean (Full Range); unit: weeks
Arm/Group | Folic Acid Supplementation | No Supplementation
Number analyzed (Participants) | 2 | 6
weeks | 4 [2 to 6] | 3.4 [2 to 8]

3. Secondary Outcome: The Number of Participants Who Developed Decreased Hemoglobin by ≥ 1 g/dl Relative to Baseline
Description: To evaluate the effect of olaparib on hemoglobin level in both arms of the study as compared to baseline before the beginning of the olaparib treatment
Time Frame: Hemoglobin levels were measured in each enrolled subject: at baseline, then every 2 weeks X 3 months, then monthly X 9 months. Accrual occurred over a 2-year period.
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid | No Supplementation
Number analyzed (Participants) | 2 | 7
Participants | 1 | 2

4. Secondary Outcome: Serum Folate
Description: To evaluate the effect of folic acid supplementation on serum folate levels as compared to the no Folate supplementation arm. Serum folate was measured every 2 weeks for the first 3 months, and then monthly for 9 months during olaparib therapy.
Time Frame: as for outcome 1
Population: We calculated the average folate level for each data point in each arm of the study.
Measure: Mean (Full Range); unit: ng/ml
Groups:
- Folic Acid Supplementation Arm: Folic Acid supplement 1 mg by mouth daily
  Folic Acid Tablet: Folic Acid 1 mg by mouth daily
Arm/Group | Folic Acid Supplementation Arm | No Supplementation
Number analyzed (Participants) | 2 | 7
ng/ml
  2 week: number analyzed (Participants) | 2 | 5
  2 week | 5.5 [3.6 to 7.3] | 7.7 [2.5 to 16.2]
  4 week: number analyzed (Participants) | 2 | 6
  4 week | 6.5 [5.5 to 21.5] | 4.6 [2.0 to 9.2]
  6 week: number analyzed (Participants) | 2 | 5
  6 week | 8.4 [7.5 to 9.3] | 7.8 [5.4 to 13.8]
  8 week: number analyzed (Participants) | 1 | 5
  8 week | 3.6 [3.6 to 3.6] | 4.0 [1.7 to 6.7]
  10 week: number analyzed (Participants) | 1 | 5
  10 week | 15.9 [15.9 to 15.9] | 8.1 [1.6 to 11.2]
  12 week: number analyzed (Participants) | 2 | 3
  12 week | 24.1 [9.6 to 38.6] | 6.1 [4.2 to 7.6]
  14 weeks: number analyzed (Participants) | 1 | 3
  14 weeks | 24.0 [24.0 to 24.0] | 10.5 [6.6 to 13.7]
  5 month: number analyzed (Participants) | 2 | 4
  5 month | 18.5 [8.3 to 28.7] | 9.5 [3.7 to 18.4]
  6 month | 11.2 [3.8 to 18.7] | 5.6 [2.8 to 8.9]
  7 month: number analyzed (Participants) | 2 | 3
  7 month | 10.5 [9.3 to 10.8] | 6.8 [5.0 to 8.8]
  8 month: number analyzed (Participants) | 2 | 2
  8 month | 13.6 [10.5 to 16.7] | 5.8 [5.5 to 6.1]
  9 month: number analyzed (Participants) | 1 | 1
  9 month | 9.1 [9.1 to 9.1] | 8.2 [8.2 to 8.2]
  10 month: number analyzed (Participants) | 2 | 1
  10 month | 11.6 [8.5 to 14.7] | 7.5 [7.5 to 7.5]
  11 month: number analyzed (Participants) | 2 | 2
  11 month | 5.9 [5.1 to 6.6] | 6.8 [4.3 to 9.3]
  12 month: number analyzed (Participants) | 1 | 2
  12 month | 12.4 [12.4 to 12.4] | 9.3 [4.5 to 14.1]
  30 day follow up: number analyzed (Participants) | 2 | 4
  30 day follow up | 6.0 [5.2 to 6.5] | 9.3 [3.2 to 16.2]

5. Secondary Outcome: Number of Participants Requiring Blood Transfusions
Description: The number of patients requiring blood transfusions during olaparib treatment was counted.
Time Frame: Over 12 months while on olaparib therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid | No Supplementation
Number analyzed (Participants) | 2 | 7
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Requiring Olaparib Dose Interruptions
Description: The number of subjects requiring interruptions in olaparib treatment for any reason was counted.
Time Frame: Over 12 months while on olaparib therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid | No Supplementation
Number analyzed (Participants) | 2 | 7
Participants | 1 | 0

7. Secondary Outcome: Number of Participants Requiring Olaparib Dose Reductions for Any Reason
Description: The number of participants requiring olaparib dose reductions for any reason was counted.
Time Frame: Over 12 months while on olaparib therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid | No Supplementation
Number analyzed (Participants) | 2 | 7
Participants | 0 | 2

8. Secondary Outcome: Number of Participants Requiring Olaparib Discontinuation
Description: The number of subjects who had their olaparib treatment discontinued was counted.
Time Frame: Over 12 months while on olaparib therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid | No Supplementation
Number analyzed (Participants) | 2 | 7
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events of olaparib therapy were collected for active participants from a range of 3 - 12 months.
Description: Adverse effects were measured using CTCAE v4.0
Arm/Group | Folic Acid | No Supplementation
All-Cause Mortality (participants affected / at risk) | 0/2 | 2/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 0/2 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Folic Acid (N=2) | No Supplementation (N=7)
FATIGUE (General disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Low accrual at a single center led to a small sample size.
2. Close serum folate monitoring with early intervention for folate deficiency could have prevented more severe anemia, blood transfusions, and olaparib dose reductions.
3. Subjects were not blinded to results and may have altered their behavior. They were encouraged to hold folate-containing multivitamins but were not required to.
4. Olaparib-induced nausea and poor oral intake could have contributed to folate deficiency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04024254/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT04024254/ICF_002.pdf